CLINICAL TRIAL: NCT05904665
Title: Circulating Tumor DNA Methylation Guided Postoperative Follow-up Strategy for Non-metastatic Colorectal Cancer: a Multicenter, Prospective, Randomized Controlled Cohort Study (FIND Trial)
Brief Title: Circulating Tumor DNA Methylation Guided Postoperative Follow-up Strategy for Non-metastatic Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junjie Peng, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FIND Trial
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Non-metastatic Colorectal Cancer; Circulating Tumor DNA Methylation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ctDNA dynamic monitoring + routine postoperative follow-up (Experimental): Dynamic monitoring of ctDNA + routine postoperative follow-up: ctDNA detection is performed within one month before surgery, within one month after surgery, and every three months after surgery, for a period of 2 years. At the same time, routine postoperative follow-up is given.
  Follow-up intervention*: After completion of adjuvant chemotherapy in the patient, if ctDNA detection suggests positive, immediate chest, abdomen, and pelvis CT and other imaging examinations are performed to determine whether there is recurrence or metastasis. If it is not confirmed, repeat imaging examinations are carried out every two months in the follow-up process, and ctDNA detection is continued every three months according to the schedule. If two consecutive ctDNA retests are negative, the above imaging follow-up will resume at the frequency of routine follow-up.
  Interventions: Diagnostic Test: ctDNA methylation dynamic monitoring
- Routine postoperative follow-up (No Intervention): Routine postoperative follow-up: Only routine postoperative follow-up is given as follows: Physical examination and CEA were performed every 3-6 months for the first 2 years, every 6 months within the third to fifth year, and then annually. Chest/abdominal/pelvis computed tomography was performed annually for up to 5 years, and colonoscopy was performed for proper patients the first year after treatment and repeated in the third year if no advanced adenoma was found and then every 5 years.

INTERVENTIONS:
Diagnostic Test: ctDNA methylation dynamic monitoring — ctDNA methylation detection is performed within one month before surgery, within one month after surgery, and every three months after surgery, for a period of 2 years.
  Arms: ctDNA dynamic monitoring + routine postoperative follow-up

SUMMARY:
Colorectal cancer (CRC) is one of the most common gastrointestinal tumors. According to the latest cancer report, the incidence and mortality rates of CRC are both ranked top 5 among malignant tumors worldwide and continue to rise. Patients who receive treatment in the early stage (stage I) have a 5-year survival rate of approximately 90%. However, for high-risk stage II and III colorectal cancer patients, the 5-year survival rate is only 40%-70%, and almost half of the patients experience postoperative recurrence and metastasis.

Circulating tumor DNA (ctDNA) is a small fraction of total cell-free DNA (cfDNA) in peripheral blood circulation, carrying tumor-specific genetic and epigenetic information. It can usually be detected in the serum or plasma of tumor patients in peripheral blood. Studies have shown that methylation detection of plasma ctDNA can be used for predicting the efficacy and prognosis of tumor postoperatively, as well as for dynamic monitoring.

Current methods for monitoring CRC recurrence include testing for carcinoembryonic antigen (CEA) in blood and periodic computed tomography (CT) scans. However, due to the low sensitivity of CEA and the radiation and cost limitations of CT examination, the disease status of postoperative CRC patients cannot be well-monitored.

ctDNA is a promising biomarker for monitoring the recurrence and metastasis of CRC. Research results have shown that ctDNA can be detected in nearly all subjects before surgery, and the changes in ctDNA levels are related to the extent of surgical resection. The detection of ctDNA after surgery generally indicates recurrence within one year. ctDNA may be a more reliable and sensitive indicator than the current standard biomarker CEA, providing a window for early intervention.

This multicenter, prospective, and randomized controlled cohort study uses a single-tube methylation-specific quantitative PCR (mqMSP) detection, which detects 10 different methylation markers and can quantitatively analyze plasma samples containing tumor DNA as low as 0.01%. This study will use the ctDNA methylation detection technology to conduct quantitative detection of ctDNA methylation in the plasma of enrolled patients, hoping to predict the recurrence and metastasis risk of patients at an earlier stage through ctDNA changes, and to explore the value of ctDNA detection in guiding postoperative follow-up for non-metastatic CRC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, regardless of gender;
2. Personal status (PS) score as over 80 or Eastern Cooperative Oncology Group (ECOG) score as 0 ~ 2;
3. Preoperative imaging examinations reveal no definite distant metastatic lesions, and postoperative pTNM staging confirms patients with stage I to III colorectal cancer;
4. Radical operation performed ;
5. With expected survival of more than 12 months;
6. The subjects (or their legal representative / Guardian) must sign the informed consent form, indicating that they understand the purpose of the study, understand the necessary procedures of the study, and are willing to participate in the study.

Exclusion Criteria:

1. Blood transfusion performed during operation or within 2 weeks before operation;
2. Incomplete baseline samples, including preoperative plasma samples;
3. Two consecutive test points missing or three plasma samples missing in total before a positive ctDNA time point;
4. Pregnant or lactating women who have fertility and do not take adequate contraceptive measures;
5. Have a history of other malignant tumors within 5 years, except cured cervical carcinoma in situ or non melanoma skin cancer;
6. Primary brain tumor or central nerve metastasis is not under control, with obvious intracranial hypertension or neuropsychiatric symptoms;
7. Patients with the following serious or uncontrollable diseases: severe heart disease, the condition is still unstable after treatment, including myocardial infarction, congestive heart failure, unstable angina pectoris, pericardial effusion with obvious symptoms or unstable arrhythmia within 6 months before enrollment; definite neuropathy or psychosis, including dementia or seizures; severe or uncontrolled infection; active disseminated intravascular coagulation and obvious bleeding tendency;
8. Significant impairment of important organ function;
9. Other conditions in which the investigator believes that the patient should not participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Secondary curative-intent rate | Up to 24 months
  This study primarily evaluates whether ctDNA-informed surveillance after surgery increases the proportion of patients with CRC recurrence who receive curative-intent or metastasis-directed therapy, compared to the standard follow-up protocol within 2 years of initial surgery.

SECONDARY OUTCOMES:
TTCR | Up to 60 months
  To exam whether ctDNA-guided surveillance leads to a reduced time to clinical recurrence (TTCR) compared to standard surveillance.
DFS | Up to 60 months
  To investigate ctDNA-based disease-free survival (ctDNA-DFS), CT-based disease-free survival (CT-DFS), and the difference between ctDNA-DFS and CT-DFS (△-DFS).
Sensitivity of postoperative ctDNA monitoring for detecting recurrence | Up to 60 months
  To investigate sensitivity of postoperative ctDNA monitoring for detecting recurrence (Sensitivity=Number of ctDNA-positive patients confirmed with recurrence by imaging/Total number of patients confirmed with recurrence by imaging).
Specificity of postoperative ctDNA monitoring for detecting recurrence | Up to 60 months
  To investigate specificity of postoperative ctDNA monitoring for detecting recurrence (Specificity= Number of ctDNA-negative patients confirmed without recurrence by imaging /Total number of patients confirmed without recurrence by imaging).
OS | Up to 60 months
  To exam whether 3- and 5-year overall survival (OS) with ctDNA-guided surveillance is comparable to that achieved with standard CT-based monitoring.
Patient-reported outcomes (quality of life) | Up to 60 months
  To assess patient-reported outcomes-quality of life (EORTC QLQ-C30)-in those receiving ctDNA-guided versus standard surveillance.
Patient-reported outcomes (fear of cancer recurrence) | Up to 60 months
  To assess patient-reported outcomes-fear of cancer recurrence (FCRI)-in those receiving ctDNA-guided versus standard surveillance.
Patient-reported outcomes (cancer-related distress) | Up to 60 months
  To assess patient-reported outcomes-cancer-related distress (IES-C)-in those receiving ctDNA-guided versus standard surveillance.
Patient-reported outcomes [emotional distress (PHQ-9 scales)] | Up to 60 months
  To assess patient-reported outcomes-emotional distress (PHQ-9 scales)-in those receiving ctDNA-guided versus standard surveillance.
Patient-reported outcomes [emotional distress (GAD-7 scales)] | Up to 60 months
  To assess patient-reported outcomes-emotional distress (GAD-7 scales)-in those receiving ctDNA-guided versus standard surveillance.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China